CLINICAL TRIAL: NCT04214275
Title: The Effect of Pulmonary Rehabilitation on Respiratory Functions and Quality of Life Following Coronial Artery Bypass Grafting: a Randomized Controlled Trial
Brief Title: Pulmonary Rehabilitation and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeliz Ciğerci, Director, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016/806
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Bypass Graft
Keywords: coronary artery bypass; pulmonary rehabilitation; quality of life; respiratory functions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): standard care and participated in a pulmonary rehabilitation program
  Interventions: Other: pulmonary rehabilitation
- control group (No Intervention): received standard care after coronary artery bypass graft

INTERVENTIONS:
Other: pulmonary rehabilitation — Simple breathing techniques, secretion-removal techniques, airway-cleaning techniques, mobilization techniques and use of an incentive spirometer
  Arms: intervention group

SUMMARY:
In this study, the effect of a pulmonary rehabilitation (PR) program on the respiratory function and quality of life of patients undergoing CABG surgery with an open-heart technique is examined. A randomized controlled experimental design was used. The study was conducted with two groups: the intervention group (n=25) and control group (n=25). The control group received standard care after CABG. In contrast, the experimental group, in addition to standard care, participated in a PR program created by the researchers. After CABG, the respiratory functions of both groups (clinical care day 4) and quality of life (6th week) evaluated

ELIGIBILITY:
Inclusion Criteria:

* Patients who were extubated in twenty-four hours,
* aged 18 or above,
* had undergone CABG surgery using the open-heart method and using a saphenous vein graft for CABG,
* who were conscious,
* without visual and hearing problems,
* who spoke Turkish,
* had not orthopedic, psychiatric and neurological problems,
* no co-morbid lung disease,
* who had not been re-operated on,
* had not postoperative cardiac dysfunction,
* had not developed postoperative atrial fibrillation,
* who were willing to participate in the study.

Exclusion Criteria:

* Patients who were not extubated in twenty-four hours,
* who were under 18 years of age,
* had not undergone CABG surgery using the open-heart method and using a saphenous vein graft for CABG,
* who were not conscious,
* were visual and hearing problems,
* who don't spoke Turkish,
* had orthopedic, psychiatric and neurological problems,
* co-morbid lung disease,
* who had been re-operated on,
* had postoperative cardiac dysfunction,
* had developed postoperative atrial fibrillation,
* who were not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
The Pulmonary Function Test (PFT) | Preoperative day
  A diagnostic criterion used to identify patients with or at risk of pulmonary dysfunction. The PFT assessment was performed using the NDD Easy on-PC spirometer. During this test, challenging expiratory volume (FEV1 % (>80)), challenging vital capacity (FVC % (>80)), FEV1/FVC ( %, >80) ratio, and Peak Expiratory air pressure (PEF % (>100)) were measured in the first second. The PFT was performed in the Chest Diseases Outpatient Clinic of the hospital preoperatively.
The Pulmonary Function Test (PFT) Change | 4th day of clinical care
  A diagnostic criterion used to identify patients with or at risk of pulmonary dysfunction. The PFT assessment was performed using the NDD Easy on-PC spirometer. During this test, challenging expiratory volume (FEV1 % (>80)), challenging vital capacity (FVC % (>80)), FEV1/FVC ( %, >80) ratio, and Peak Expiratory air pressure (PEF % (>100)) were measured in the first second. The PFT was performed in the Chest Diseases Outpatient Clinic of the hospital preoperatively. The PFT was performed in the Chest Diseases Outpatient Clinic of the 4th day of clinical care.

SECONDARY OUTCOMES:
The Short-Form Health Survey (SF-36) | preoperative day
  The points given vary between 0-100; 0 points indicate bad health and 100 points indicate that health is progressing in a good direction.
The Short-Form Health Survey (SF-36) Change | postoperative sixth week
  The points given vary between 0-100; 0 points indicate bad health and 100 points indicate that health is progressing in a good direction.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Ciğerci, PhD, Principal Investigator — +90 272 444 0304
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes